CLINICAL TRIAL: NCT07157124
Title: A Theory-Informed Examination of a Brief Visuospatial Intervention and Its Mechanisms for Reducing Alcohol Cravings and Consumption
Brief Title: Examining the Effectiveness of Dynamic Visual Noise (DVN) for Reducing Alcohol Cravings and Consumption in College Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wyoming (Other)
Responsible Party: Principal Investigator, Emma Winterlind, Clinical Psychology Doctoral Student, University of Wyoming
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-2025-162
Record Dates: First submitted 2025-08-21; First posted 2025-09-05 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Craving; Alcohol Drinking
Keywords: alcohol craving; dynamic visual noise; alcohol consumption; attentional bias; craving; alcohol; DVN; static visual noise; SVN
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: Participants will be block randomized by sex into one of the two arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic Visual Noise (DVN) (Experimental)
  Interventions: Other: Dynamic Visual Noise (DVN)
- Static Visual Noise (SVN) (Sham Comparator)
  Interventions: Other: Static Visual Noise (SVN)

INTERVENTIONS:
Other: Dynamic Visual Noise (DVN) — DVN is a brief visual array of patterns of flickering black and white dots. In alignment with prior literature, the DVN array will consist of an 80 x 80 grid of 4 x 4 black and white pixel squares that will change at a rate of 640 frames per second. The DVN will be 30 seconds in duration, though participants will be able to keep watching for as long as desired by restarting the video of the array.
  Arms: Dynamic Visual Noise (DVN)
Other: Static Visual Noise (SVN) — SVN is similar to DVN, but refers to a static (or still) image of an array of black and white squares. The SVN will consist of an 80 x 80 grid of 4 x 4 black and white pixel squares. SVN has been used in previous working memory-loading studies as a control for DVN. Similar to the DVN, participants in the control group will view the SVN for at least 30 seconds (but they will be able to keep viewing it for as long as desired).
  Arms: Static Visual Noise (SVN)

SUMMARY:
The goal of this clinical trial is to examine whether dynamic visual noise (DVN), a short video array of rapidly moving black and white squares, reduces cravings for and consumption of alcohol in college students who drink alcohol and experience cravings for alcohol at least once a week on average. A second goal of this clinical trial is to examine whether changes in attentional bias towards alcohol (that is, the tendency to pay greater mental and visual attention towards alcohol over other things in one's environment) is a mechanism by which DVN reduces alcohol cravings and consumption.

Researchers will compare DVN to static visual noise (SVN), which is a still image of black and white squares that has been used as a control condition for DVN in prior literature.

Participants will:

1. Visit the laboratory once to complete the baseline data collection
2. Watch the DVN or SVN every day for seven days (including the day of the laboratory visit)
3. Complete daily follow-ups for six days following the day of the laboratory visit
4. Complete a final follow-up on the seventh day following the laboratory visit

ELIGIBILITY:
Inclusion Criteria:

1. Must report being between the age of 18 and 29
2. Must report drinking alcohol at least once per week on average over the past month
3. Must report having drank beer or alcoholic seltzers in the past month
4. Must endorse experiencing craving at least once per week over the past month, on average
5. Must report not currently receiving nor planning to seek any other treatment for their alcohol use within the next 30 days
6. Must report owning a personal electronic device with access to the Internet
7. Must report owning or having access to a computer with access to the Internet

Exclusion Criteria:

1. Major visual impairment (i.e., legal blindness or color blindness)
2. History of seizures and/or diagnosed seizure disorder
3. Current medical diagnosis provided by a qualified professional (i.e., psychologist, psychiatrist, neurologist) that is characterized by cognitive impairment (i.e., neurocognitive disorder due to traumatic brain injury, traumatic brain injury, HIV infection, post-concussive syndrome, and intellectual disability)
4. Concussion in the past month
5. A current diagnosis of any substance use disorder besides alcohol use disorder, as determined by a qualified professional (i.e., psychologist, psychiatrist)

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Strength of Alcohol Craving | Baseline and 1-week follow-up
  Strength of alcohol craving will be measured using the Craving Experiences Questionnaire - Strength (CEQ-S). The measure inquires about the individual's past-week craving experiences. Higher average scores indicate stronger past-week cravings. Changes in mean craving will be calculated as changes in mean strength of past-week alcohol craving at follow-up relative to baseline for each condition.
Frequency of Craving | Baseline and 1-week follow-up
  Frequency of alcohol craving will be measured using the Craving Experiences Questionnaire - Frequency (CEQ-F). The measure inquires about the individual's past-week craving experiences. Higher average scores indicate more frequent past-week craving. Changes will be calculated as changes in mean frequency of past-week alcohol craving at follow-up relative to baseline for each condition.
Alcohol Consumption | Baseline and 1-week follow-up
  At baseline and follow-up, participants will complete the Daily Drinking Questionnaire (DDQ) to indicate the extent of their past-week alcohol consumption. Higher total scores indicate more past-week alcohol consumption. Changes will be calculated as changes in mean past-week alcohol use at follow-up relative to baseline for each condition.
Attentional Bias towards Alcohol | Baseline and 1-week follow-up
  Attentional bias will be measured at the initial laboratory session and at the 1-week final follow-up via the Alcohol Visual Probe task. Changes will be examined as mean changes in reaction time at follow-up minus reaction time at baseline for each condition.

SECONDARY OUTCOMES:
Immediate Changes in Strength of Alcohol Craving Before and After DVN/SVN Task | Baseline
  Participants will view their assigned intervention (i.e., DVN or SVN) as part of the initial baseline visit. Participants will first undergo a craving induction paradigm. Participants will then complete the CEQ-Strength-Now (CEQ-S-N) to indicate the strength of their current craving. Then, participants will view the DVN or SVN (depending on their assigned condition). After viewing the task, participants will complete the CEQ-S-N again. Higher average scores on the CEQ-S-N indicate stronger current moment cravings. Immediate changes in craving will be calculated as the average CEQ-S-N score before viewing the task minus average CEQ-S-N score after viewing the task. A mean change score will be calculated for each condition.
Immediate Changes in Strength of Craving Before and After DVN/SVN | 1-Week Intervention Period, Between Baseline Visit and 1-week Follow-Up
  During the intervention phase, participants will be able to freely access their assigned intervention whenever they experience a craving. When they access the intervention, participants will first be asked to indicate, using a 0-100 Visual Analogue Scale (VAS), the strength of their current cravings for alcohol (i.e., "How strong is your craving for alcohol RIGHT NOW?"). They will then view their assigned intervention for at least 30 seconds. Immediately after viewing their intervention, they will complete the same VAS item. The change score will be calculated as the craving score before viewing minus the craving score after each viewing. A mean change score will be calculated for each condition.

OTHER OUTCOMES:
Changes in Negative Affect from Baseline to Final Follow-Up | Baseline and 1-week follow-up
  Negative affect (NA) is proposed to be an associative stimulus that may elicit cravings under the Elaborated Intrusion theory. However, DVN has never been examined in the context of affect. As such, the one and only exploratory aim of the study is to examine whether DVN affects NA, longitudinally and/or immediately. NA will be measured through the use of the NA subscale of the Positive and Negative Affect Schedule (PANAS) at baseline and final follow-up. Changes will be calculated as changes in mean NA at follow-up relative to baseline. Mean change scores will be calculated for each condition.
Changes in Negative Affect Immediately after Viewing DVN/SVN | Baseline
  Negative affect (NA) is proposed to be an associative stimulus that may elicit cravings under the Elaborated Intrusion theory. However, DVN has never been examined in the context of affect. As such, the one and only exploratory aim of the study is to examine whether DVN affects NA, longitudinally and/or immediately. NA will be measured through the use of the NA subscale of the Positive and Negative Affect Schedule (PANAS). Participants will complete the measure immediately before and after viewing the DVN/SVN during their baseline session. Changes in NA will be calculated as average NA score after viewing minus average NA score before viewing. Mean change scores will be calculated for each condition.
Past-year Alcohol Use Severity | Baseline
  To characterize and describe the sample in terms of their alcohol use and related experiences, participants will complete the Alcohol Symptom Checklist (ASC), a measure of alcohol use severity wherein each item corresponds to a diagnostic criteria of alcohol use disorder outlined in the Diagnostic and Statistical Manual of Mental Disorders 5th edition. Higher total scores indicate more severe past-year alcohol use. Mean scores will be calculated for each condition.
Past-month Negative Alcohol Consequences | Baseline
  To characterize and describe the sample in terms of their alcohol use and related experiences, participants will complete the Brief Young Adult Alcohol Consequences Questionnaire (B-YAACQ) at baseline. Higher total scores indicate more negative alcohol consequences experienced in the past month. Mean scores will be calculated for each condition.
Past-month Alcohol Use | Baseline
  To characterize and describe the sample in terms of their alcohol use and related experiences, participants will complete the DDQ for their past-month alcohol use at baseline. Higher total scores indicate greater quantity and frequency of alcohol use. Mean past-month alcohol use will be calculated for each condition.
Attention Validation | 1-Week Intervention Period, Between Baseline Visit and 1-week Follow-Up
  During the intervention period, participants will have free access to their assigned intervention. After they view the intervention, they will be asked two questions regarding the extent to which they paid attention to the intervention. Questions will include:
  1. How many times did you look away from the task, even if only for a brief moment?
  2. If you looked away at any point, approximately how long did you look away for in total? (Participants select a response option between "N/A; I did not look away" to 15+ seconds).
  Average number of times and average duration of looking away will be calculated for each condition.
Number of Times Intervention was Viewed / Acceptability & Feasibility | 1-Week Intervention Period, Between Baseline Visit and 1-week Follow-Up
  During the intervention period, participants will have free access to their assigned intervention and be instructed to view it at least once per day but ideally any time they experience a craving. The average number of times the intervention was accessed will be calculated for each condition as an indicator of acceptability and feasibility.
Daily Alcohol Consumption | 1-Week Intervention Period, Between Baseline Visit and 1-week Follow-Up
  We will be gathering data on whether participants have consumed alcohol that day, when the most recent time they consumed alcohol was, and whether they are currently under the influence of alcohol. After participants finish viewing their assigned task, answer questions about their current craving, and answer the attention validation items, they will answer the following questions about their recent alcohol use:
  1. Have you consumed any alcohol since the last time you completed this task?
  2. Approximately, how many hours has it been since your last alcoholic drink (round to the closest hour)?
  3. Are you currently experiencing any effects of alcohol? That is, have you recently consumed alcohol and are experiencing alcohol intoxication (i.e., feeling "tipsy" or "drunk"?)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wyoming, Laramie, Wyoming, United States

IPD SHARING:
Plan to Share IPD: No